CLINICAL TRIAL: NCT03956173
Title: Hypoglycemia and Cardiac Arrhythmias in Type 1 Diabetes
Acronym: Hypo-Heart-1
Status: Completed | Type: Observational
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Hillerod Hospital, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: H-18034040
Record Dates: First submitted 2018-10-12; First posted 2019-05-20 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2022-07

CONDITIONS: Diabetes type1; Hypoglycemia; Arrhythmias, Cardiac
MeSH Terms: conditions — Hypoglycemia; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clamp group: 24 patients with type 1 diabetes.
  Interventions: Other: Hypoglycemic combined with either normo or hyperglycemic clamp.

INTERVENTIONS:
Other: Hypoglycemic combined with either normo or hyperglycemic clamp. — Twenty-four patients with type 1 diabetes has been recruited for a cross-over study including two experimental days, a combined hypo- and hyperglyemic clamp and a combined hypo- and euglycemic clamp, respectively. Patients will be randomised 1:1 to start with either the combined hypo- and hyperglycemic or the hypo- and euglycemic clamp. The hypo- and hyperglycemic or the hypo- and euglycemic clamp are estimated to last 255 minutes. The two clamp days will be separated by at least 30 days.

SUMMARY:
The investigators hypothesise that following episodes of hypoglycemia, rebound hyperglycemia may result in a prolonged period of increased QTc and, thereby, increased susceptibility to serious cardiac arrhythmias in patients with type - 1 diabetes.

DETAILED DESCRIPTION:
In this study, changes in cardiac rhythm, haemodynamic regulation, and hormonal response will be evaluated during insulin-induced hypoglycemia followed by hyperglycemia and euglycemia, respectively, on two separate experimental days. Twenty-four patients with type-1 diabetes are included. Patients are randomised 1:1 to start with either the combined hypo- and hyperglycemic or the hypo- and euglycemic clamp. After an overnight 10 hour fast, participants are admitted for a 255 minute clamp. An individualised insulin infusion will be initiated targeting a plasma glucose level of 5.0-8.0 mmol/l. When the targeted plasma glucose level is achieved, the hyperinsulinemic euglycemic clamp will be initiated at time 0. The insulin infusion will be fixed at an infusion rate 80 mU/m2/min and a 20% glucose infusion will be initiated in order to regulate plasma glucose levels. After 45 min of monitoring at euglycemic plasma glucose level, plasma glucose will be decreased over a period of 30 minutes, targeting 2.5 mmol/l for a period of 60 min in a hyperinsulinemic hypoglycemic clamp. From 135 min to 195 min, plasma glucose levels will be increased to either hyperglycemic level or euglycemic level and will be kept constant for 105 minutes. Echocardiography is performed at baseline, at hypoglycemic level and at hyper-or normoglycemic level. Blood samples are taken every 15 minutes throughout the entire clamp, however bedside plasma glucose is analysed every fifth minute. A Holter-ECG is obtained throughout the entire clamp.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent
* Type 1 diabetes diagnosed according to the criteria of the World Health Organization (WHO)
* Age 18-70 years
* Insulin treatment for ≥3 years

Exclusion Criteria:

* Arrhythmia diagnosed prior to the screening visit
* Implantable cardioverter defibrillator (ICD) or pacemaker at the time of inclusion
* Severe heart failure (left ventricular ejection fraction <25%)
* Structural heart disease (Wolf-Parkinson-White syndrome, congenital heart disease, severe valve disease)
* Thyroid dysfunction (except for well-regulated eltroxin substituted myxoedema)
* Anemia (male: hemoglobin <8.0; female: hemoglobin <7.0 mmol/l)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 24 patients with type 1 diabetes with insulin treatment for ≥ 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
QTc prolongation. | 255 minutes
  Difference in mean corrected QT interval (QTc) prolongation during hyperglycemia compared to euglycemia both preceded by insulin induced hypoglycemia

SECONDARY OUTCOMES:
QTd dispersion. | 255 minutes
  Difference in QT dispersion (QTd) during hyperglycemia compared to euglycemia both preceded by insulin induced hypoglycemia
Atrial ectopic beats. | 255 minutes
  Difference in atrial ectopic beats (prematurity threshold 30%),during hyperglycemia compared to euglycemia both preceded by insulin-induced hypoglycemia
Bradycardia | 255 minutes
  Difference in non-clinically significant bradycardia (≤45 bpm for 5 seconds) during hyperglycemia compared to euglycemia both preceded by insulin-induced hypoglycemia
Ventricular premature beats | 255 minutes
  Difference in ventricular premature beats during hyperglycaemia compared to euglycaemia both preceded by insulin-induced hypoglycaemia
Glucagon response | 255 minutes
  Differences in glucagon response during hyperglycemia compared to euglycemia both preceded by insulin induced hypoglycemia
Catecholamine response | 255 minutes
  Differences in catecholamine response during hyperglycemia compared to euglycemia both preceded by insulin induced hypoglycemia
Growth hormone response | 255 minutes
  Differences in growth hormone response during hyperglycemia compared to euglycemia both preceded by insulin induced hypoglycemia
Cortisol response | 255 minutes
  Differences in cortisol responses during hyperglycemia compared to euglycemia both preceded by insulin induced hypoglycemia
Haemodynamic regulation. | 255 minutes
  Differences in haemodynamic regulation (measured by echocardiography) during hyperglycemia compared to euglycemia both preceded by insulin-induced hypoglycemia
Inflammatory response | 255 minutes
  Differences in markers of inflammation (high-sensitive C-reactive peptide (hs-CRP) and interleukin 6 (IL-6)) during hyperglycemia compared to euglycemia both preceded by insulin-induced hypoglycemia
Oxidative stress markers (8-iso-PGF2α) | 255 minutes
  Differences in markers of oxidative stress (8-iso prostaglandin F2α (8-iso-PGF2α)) during hyperglycemia compared to euglycemia both preceded by insulin-induced hypoglycemia
Oxidative stress markers (8-oxoGuo) | 255 minutes
  Differences in markers of oxidative stress (8-oxo-7,8-dihydroguanosine (8-oxoGuo)) during hyperglycemia compared to euglycemia both preceded by insulin-induced hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Tina Vilsbøll, MD, DMSc, Study Director — Steno diabetic centre (SDCC)
Locations (1):
- Clinical Metabolic Physiology, SDCC, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided